CLINICAL TRIAL: NCT05435105
Title: The Effect of Virtual Reality and Local Cold-Vibration Methods on Reducing Anxiety, Fear and Pain Due to Peripheral Intravenous Catheterization in Children
Brief Title: Effects of Virtual Reality, Cold-Vibration Due To Intravenous Catheterization on Pain, Fear and Anxiety on Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Berfu Atalay, Nurse, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019/881; 5208 (Other: AkdenizU Scientific Research Projects Coordination Unit)
Record Dates: First submitted 2022-06-17; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Procedural Anxiety; Fear; Procedural Pain; Child, Only
Keywords: procedural anxiety; fear; procedural pain; peripheral intravenous catheter; virtual reality; local-cold vibration; distraction method; nonpharmacological method
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Intervention Model Description: A total of three groups as 2 intervention (virtual reality, local cold-vibration) and control group (routine application)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Group (Experimental): Watching the cartoon by wearing virtual reality glass to the child during the peripheral intravenous catheterization
  Interventions: Behavioral: Virtual reality
- Local Cold-Vibration Group (Experimental): The local cold-vibration device is placed 5 cm above the area just before peripheral intravenous catheterization
  Interventions: Behavioral: Local cold-vibration
- Control Group (No Intervention): Routine Care

INTERVENTIONS:
Behavioral: Virtual reality — Distraction method
  Arms: Virtual Reality Group
Behavioral: Local cold-vibration — Distraction method
  Arms: Local Cold-Vibration Group

SUMMARY:
This is a randomized controlled trial. The aim of the study is to the effects of Virtual Reality and Local Cold-Vibration applications in reducing anxiety, fear and pain due to intravenous catheterization (PIC) in children aged 5-10 years. PIC was found to be effective in reducing anxiety, fear and pain due to peripheral intravenous catheterization.

DETAILED DESCRIPTION:
Peripheral intravenous catheterization is an administration method that is frequently used in children and causes pain. There are different non-pharmacological methods for reducing pain due to invasive procedures. The use of non-pharmacological methods is an important part of nursing care to reduce the short and long-term negative effects of painful interventions on children.This study was planned to compare the effectiveness of virtual reality and local cold-vibration applications in reducing anxiety, fear and pain caused by PIC in children aged 5-10 years. It was planned as a randomized controlled experimental study in pre-test, post-test design. The sample of the study was carried out in the Pediatric Emergency Unit of Akdeniz University Medical Faculty Hospital. The applicant will consist of 120 children aged 5-10 years. There will be a total of three groups in the research, 2 of which are the intervention group (virtual reality, local cold-vibration) and the control group (routine application). Data will be collected using the "Child-Parent Description Form", "Child Anxiety Scale-State Scale", "Child Fear Scale", "Wong- Baker Faces Pain Scale". Data will be collected before and within the first 5 minutes after IM injection administration. Scales; to be filled in separately by the child, one of the parents, and the nurse administering the PIC. As a result of this study, it was concluded that the use of virtual reality glasses and local cold-vibration methods are effective in reducing the pain, anxiety and fear that due to PIC placement in children aged 5-10 years.

ELIGIBILITY:
Inclusion Criteria:

the child;

* between the ages of 5-10
* PIC application will be made
* No visual, auditory or sensory loss
* Mental and language deficiencies
* Those who have not taken any analgesic medication in the last 4 hours
* Do not have a chronic disease (such as oncological diseases, chronic kidney failure) that causes repeated admissions or hospitalizations to the hospital.

Exclusion Criteria:

* Unsuccessful PIC application in the first time
* The child in the group with local cold-vibration application removes the device during the procedure (PIC application).
* The child in the group in which virtual reality was applied, removing the virtual reality glasses during the procedure (PIC application).
* Suspecting 'Covid 19' (having any of the symptoms such as fever, cough, respiratory distress, chest pain, loss of taste and smell, sore throat)

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2022-06-27 (Estimated)

PRIMARY OUTCOMES:
Assessing the children's anxiety with Children's State Anxiety | Before the peripheral intravenous catheterization
  The Children's State Anxiety (CAS-S). The CAS-S assesses children's anxiety and uses before medical procedures. This scale is drawn like a thermometer with a bulb at the bottom and also includes horizontal lines at intervals going up to the top (0-10). This scale ranges from 0 to 10. Higher values represent higher anxiety
Assessing the children's anxiety with Children's State Anxiety | Within the first 5 minutes after the peripheral intravenous catheterization
  The Children's State Anxiety (CAS-S). The CAS-S assesses children's anxiety and uses before medical procedures. This scale is drawn like a thermometer with a bulb at the bottom and also includes horizontal lines at intervals going up to the top (0-10). This scale ranges from 0 to 10. Higher values represent higher anxiety
Assessing the children's fear with Child Fear Scale | Before the peripheral intravenous catheterization
  The Child Fear Scale (CFS). The Child Fear Scale will use.This one-item scale measures procedure-related fear in children, consists of five sex-neutral faces, ranges from 0 (no fear) to extreme fear. This rating scale ranges from 0 to 4. It ranges from a no fear (neutral) face (0) on the far left to a face showing extreme fear on the far right. Higher scores mean a worse outcome. The rater responds indicates the level of fear.
Assessing the children's fear with Child Fear Scale | Within the first 5 minutes after the peripheral intravenous catheterization
  The Child Fear Scale (CFS). The Child Fear Scale will use.This one-item scale measures procedure-related fear in children, consists of five sex-neutral faces, ranges from 0 (no fear) to extreme fear. This rating scale ranges from 0 to 4. It ranges from a no fear (neutral) face (0) on the far left to a face showing extreme fear on the far right. Higher scores mean a worse outcome. The rater responds indicates the level of fear.
Assessing the children's pain with Wong-Baker-FACES | Before the peripheral intravenous catheterization
  Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10. Faces show emotions from smiling (0 = very happy/ no pain) to crying (10 = hurts worst).
Assessing children's pain with Wong-Baker-FACES | Within the first 5 minutes after the peripheral intravenous catheterization
  Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10. Faces show emotions from smiling (0 = very happy/ no pain) to crying (10 = hurts worst).

CONTACTS AND LOCATIONS:
Overall Officials: AYŞEGÜL İŞLER DALGIÇ, Professor, Study Director — Akdeniz University
Locations (1):
- Ayşegül İşler Dalgiç, Antalya, Akdeniz University, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No